CLINICAL TRIAL: NCT04513522
Title: A Phase 4 Study of Nivolumab in Combination With Ipilimumab in Patients With Previously Untreated Advanced Renal Cell Carcinoma and Intermediate-or Poor-risk Factors Conducted in India
Brief Title: A Study to Evaluate the Safety and Efficacy of Nivolumab With Ipilimumab in Participants With Untreated Advanced Kidney Cancer Conducted in India
Acronym: CheckMate 7C9
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA209-7C9
Record Dates: First submitted 2020-08-13; First posted 2020-08-14 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Kidney Neoplasms
MeSH Terms: conditions — Kidney Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Nivolumab + ipilimumab (Experimental)
  Interventions: Biological: Nivolumab; Biological: Ipilimumab

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558; Opdivo
Biological: Ipilimumab — Specified dose on specified days
  Other Names: BMS-734016; Yervoy

SUMMARY:
The purpose of this study is to assess the safety and efficacy of nivolumab combined with ipilimumab in intermediate and poor-risk participants with previously untreated advanced renal cell carcinoma (RCC) or metastatic RCC (mRCC) in India.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmation of renal cell carcinoma (RCC) with clear cell component including participants who may have sarcomatoid features
* Qualifies as intermediate or poor risk by meeting at least one of the prognostic factors as per the International Metastatic RCC Database Consortium (IMDC) criteria
* Indian participants with Indian ethnicity living in India
* No prior systemic therapy for RCC
* Measurable disease lesion by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria

Exclusion Criteria:

* Participants with active, untreated, symptomatic central nervous system (CNS) metastases
* Major surgery less than 28 days prior to the first dose of study treatment
* Participants with an autoimmune disease, or any other condition, requiring systemic treatment with either corticosteroids or other immunosuppressive medications

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (11):
- India (11):
  - Local Institution - 0005, Ahmedabad, Gujarat
  - Local Institution - 0011, Trivandrum, Kerala
  - Local Institution - 0013, Mumbai, Maharashtra
  - Local Institution - 0001, Mumbai, Maharashtra
  - Local Institution - 0007, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0006, Bangalore
  - Local Institution - 0017, Delhi
  - Local Institution - 0002, Karnataka
  - Local Institution - 0019, Kolkata
  - Local Institution - 0016, Mumbai
  - Local Institution - 0012, Pune

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + Ipilimumab: Participants received nivolumab 3mg/kg Q3W combined with ipilimumab 1mg/kg Q3W for 4 doses followed by nivolumab 3mg/kg Q2W for up to 52 weeks.
Period: Overall Study
Arm/Group | Nivolumab + Ipilimumab
Started | 101
Completed | 36
Not Completed | 65
Not completed — Other reasons | 1
Not completed — Adverse event unrelated to study drug | 9
Not completed — Study drug toxicity | 14
Not completed — Disease progression | 39
Not completed — Participants withdrew consent | 2

BASELINE CHARACTERISTICS:
Population: All treated participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.0 (9.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 79
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian Indian | 101

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Participants Experiencing High Grade Immune-Mediated Adverse Events (IMAE)
Description: IMAEs are a type of adverse event that occurs when the immune system reacts against the body's own tissues, including diarrhea/colitis, hepatitis, pneumonitis, nephritis and renal dysfunction, rash, and endocrine (adrenal insufficiency, hypophysitis, hypothyroidism/thyroiditis, hyperthyroidism, and diabetes mellitus). IMAE analyses includes events, regardless of causality, which occurred during the study and follow-up. Only participants who received immune-modulating medication for treatment of the event are reported, with the exception of endocrine events, which will be included regardless of treatment since these events are often managed without immunosuppression.
  High grade (Grade 3 to 4 and Grade 5) IMAEs are reported. IMAEs are graded on a scale from 1 to 5, in which Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events may require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose until 100 days after the last dose or for a maximum of 52 weeks from the date of the first on-study dose of nivolumab, whichever occurs earlier.
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 101
Participants
  Pneumonitis Grade 3-4 | 2
  Nephritis and Renal Dysfunction Grade 3-4 | 1
  Rash Grade 3-4 | 2
  Adrenal Insufficiency Grade 3-4 | 1
  Diarrhea/Colitis Grade 3-5 | 0
  Hepatitis Grade 3-5 | 0
  Nephritis and Renal Dysfunction Grade 5 | 0
  Rash Grade 5 | 0
  Hypersensitivity Grade 3-5 | 0
  Adrenal Insufficiency Grade 5 | 0
  Hypothyroidism/Thyroiditis Grade 3-5 | 0
  Diabetes Mellitus Grade 3-5 | 0
  Hyperthyroidism Grade 3-5 | 0
  Hypophysitis Grade 3-5 | 0

2. Secondary Outcome: Time to Onset of High Grade Immune-Mediated Adverse Event (IMAE)
Description: Time to onset is defined as the time between the day of the first dose of study treatment and the onset date of the earliest AE (Grades 3-5) in this category. All IMAEs that occurred between first dose and 100 days past last dose are recorded. IMAEs are a type of adverse event that occurs when the immune system reacts against the body's own tissues. IMAE analyses includes events, regardless of causality, which occurred during the study and follow-up. Only participants who received immune-modulating medication for treatment of the event are reported, with the exception of endocrine events, which will be included regardless of treatment since these events are often managed without immunosuppression.
  High grade (Grades 3 through 5) IMAEs are reported. IMAEs are graded on a scale from 1 to 5, in which Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events may require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose until onset of IMAE (up to approximately 15 months)
Population: All treated participants who experienced at least 1 IMAE
Measure: Median (Full Range); unit: Weeks
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 11
Weeks
  ADRENAL INSUFFICIENCY: number analyzed (Participants) | 1
  ADRENAL INSUFFICIENCY | 9.9 [9.9 to 9.9]
  PNEUMONITIS: number analyzed (Participants) | 2
  PNEUMONITIS | 7.29 [1.4 to 13.1]
  NEPHRITIS AND RENAL DYSFUNCTION: number analyzed (Participants) | 1
  NEPHRITIS AND RENAL DYSFUNCTION | 20.00 [20.0 to 20.0]
  RASH: number analyzed (Participants) | 2
  RASH | 29.21 [29.0 to 29.4]

3. Secondary Outcome: Time to Resolution of High Grade Immune-Mediated Adverse Event (IMAE)
Description: Time to resolution of IMAEs is defined as the longest time from onset to complete resolution or improvement to the grade at baseline among all clustered AEs experienced by the participant in this category per adverse event criteria category. Events which worsened into grade 5 events (death) or have a resolution date equal to the date of death are considered unresolved. If a clustered AE is considered as unresolved, the resolution date will be censored to the last known alive date. Improvement to the grade at baseline implies that all different events in the clustered adverse event should at least have improved to the corresponding (i.e. with same preferred term) baseline grade.
  High grade (Grades 3 through 5) IMAEs are reported. IMAEs are graded on a scale from 1 to 5, in which Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events may require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose until resolution of IMAE (up to approximately 15 months)
Population: All treated participants who experienced at least 1 IMAE that was resolved. Participants who experienced an IMAE that did not resolve were censored.
Measure: Median (Full Range); unit: Weeks
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 9
Weeks
  ADRENAL INSUFFICIENCY: number analyzed (Participants) | 1
  ADRENAL INSUFFICIENCY | 1.1 [1.1 to 1.1]
  RASH: number analyzed (Participants) | 2
  RASH | 10.07 [5.0 to 15.1]

4. Secondary Outcome: The Number of Participants Who Received Immune-Modulating Medication
Description: Immune modulating medications are medications entered on an immune modulating medication form or available from the most current pre-defined list of immune modulating medications. This list is revisited whenever UMC WHO releases a new version and updated accordingly.
Time Frame: From first dose up to 100 days after last dose (up to approximately 15 months)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 101
Participants | 38

5. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) was defined as the number of participants with a best overall response of confirmed Complete Response (CR) or Partial Response (PR) (per RECIST 1.1 criteria) divided by the number of all treated participants. RECIST 1.1 = Response Evaluation Criteria in Solid Tumors. CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose up to 100 days after last dose (up to approximately 15 months)
Population: All response evaluable participants - a total of 16 participants were excluded from "all response evaluable participants" population as they did not have measurable disease at baseline or at least 1 evaluable on-study assessment
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 85
Percentage of participants | 37.6 [27.4 to 48.8]

6. Secondary Outcome: Time to Response (TTR)
Description: TTR is defined as the time from the date of first dose to the date of the first confirmed documented response (CR or PR). For the non-responders, TTR was censored at the maximum time of response + 1 day of all participants.
  CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From first dose to the date of CR or PR (up to approximately 15 months)
Population: All confirmed responders
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 32
Months | 2.79 [2.3 to 10.3]

7. Secondary Outcome: Duration of Response (DoR)
Description: Duration of Response (DOR) is defined as the time between the date of first documented response (CR or PR) that was subsequently confirmed to the date of the first documented progression as determined using RECIST 1.1, or death due to any cause, whichever occurs first. For participants who neither progress nor die, the duration of response will be censored on the date of their last evaluable tumor assessment. For participants who start subsequent therapy before progression or die, the duration of response will be censored on the date of their last evaluable tumor assessment conducted on or prior to the initiation of the subsequent therapy.
  CR= Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Analysis based on Kaplan Meier estimates.
Time Frame: From first documented response (CR or PR) up to first documented progression or death due to any cause, whichever occurs first (up to approximately 3 years)
Population: All treated participants who have measurable disease at baseline and at least one on-study assessment
Measure: Median (Full Range); unit: Months
Arm/Group | Nivolumab + Ipilimumab
Number analyzed (Participants) | 4
Months | NA [1.3 to 9.9] — Median not calculated due to not reaching the KM 50% threshold

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their randomization to study completion, (up to approximately 3 years). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 15 months)
Arm/Group | Nivolumab + Ipilimumab
All-Cause Mortality (participants affected / at risk) | 11/101
Serious Adverse Events (participants affected / at risk) | 37/101
Other Adverse Events (participants affected / at risk) | 80/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=101)
Anaemia (Blood and lymphatic system disorders) | 3
Acute coronary syndrome (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Hyperthyroidism (Endocrine disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Death (General disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 1
Pyrexia (General disorders) | 1
Bile duct stone (Hepatobiliary disorders) | 1
Contrast media reaction (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Altered state of consciousness (Nervous system disorders) | 1
Guillain-Barre syndrome (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hemiplegia (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 2
Acquired hydrocele (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + Ipilimumab (N=101)
Anaemia (Blood and lymphatic system disorders) | 14
Hyperthyroidism (Endocrine disorders) | 10
Hypothyroidism (Endocrine disorders) | 10
Constipation (Gastrointestinal disorders) | 9
Diarrhoea (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 11
Asthenia (General disorders) | 19
Fatigue (General disorders) | 11
Pain (General disorders) | 6
Pyrexia (General disorders) | 17
Blood creatinine increased (Investigations) | 10
Weight increased (Investigations) | 6
Decreased appetite (Metabolism and nutrition disorders) | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 6
Hyponatraemia (Metabolism and nutrition disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 25
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 21
Rash (Skin and subcutaneous tissue disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT04513522/Prot_SAP_000.pdf